CLINICAL TRIAL: NCT02129049
Title: Enhancing Connections Telephone Program: A Cancer Education Program for Parents
Brief Title: Telephone-Based Educational Intervention in Improving Communication Between Patients With Stage 0-III Cancer and Their Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 9095; NCI-2014-00928 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9095 (Other: Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium); R03CA178488 (NIH); P30CA015704 (NIH)
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2016-03-09 (Estimated); Status verified 2016-03

CONDITIONS: Breast Cancer; Cervical Cancer; Colon Cancer; Leukemia; Lymphoma; Malignant Neoplasm; Melanoma; Rectal Cancer
MeSH Terms: conditions — Breast Neoplasms; Uterine Cervical Neoplasms; Colonic Neoplasms; Leukemia; Lymphoma; Neoplasms; Melanoma; Rectal Neoplasms | interventions — Early Intervention, Educational; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Supportive care (Enhancing Connections Telephone Program) (Experimental): See Detailed Description.
  Interventions: Other: educational intervention; Behavioral: telephone-based intervention; Other: questionnaire administration

INTERVENTIONS:
Other: educational intervention — Participate in the Enhancing Connections Telephone Program
  Other Names: intervention, educational
Behavioral: telephone-based intervention — Participate in the Enhancing Connections Telephone Program
Other: questionnaire administration — Ancillary studies

SUMMARY:
This pilot clinical trial studies the feasibility of a telephone-based educational intervention in improving communication between patients with stage 0-III cancer and their children. An educational program delivered by telephone may help parents talk with their school-age child about their cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Test the feasibility of the recruitment and study protocol.

II. Evaluate the short-term impact of the program on the diagnosed parents' and the parent's perceptions of their children's adjustment using a within group design (pre-posttest design).

III. To compare outcomes from the telephone-delivered program with outcomes obtained from the in-person program (between group design).

OUTLINE:

Participants complete the Enhancing Connections Telephone Program comprising 5, 1 hour educational telephone sessions over 3 months. During session 1, parents receive help defining the child's experience with the cancer as distinct from their own and ways to manage their own cancer-related emotions so that they do not emotionally flood the child. During session 2, parents receive assistance with developing skills to deeply listen and attend to the child's thoughts and feelings, complementing the parent's tendency to be a teacher, not a deep listener, of the child's thoughts, concerns, worries or understandings. During session 3, parents receive additional communication and parenting skills enabling them to initiate difficult cancer-related conversations and also interact with an upset child or one who is not forthcoming. During session 4, parents receive help focusing on and non-judgmentally interpreting the child's ways of coping with the cancer. It includes exercises that assist the parent to relinquish negative assumptions about the child's behavior related to the parent's cancer. Concurrently the session offers the ill parent ways to elicit their child's report of what the parent can do to assist the child cope with the child's cancer-related pressures. During session 5, parents focus on the gains they made in prior sessions and what they have accomplished, in their own words, in parenting their child about the cancer. The session also assists the ill parent to identify available resources that can be used after program completion to maintain the parent's newly acquired gains from the program.

ELIGIBILITY:
Inclusion Criteria:

* Parents will be eligible if they have an initial diagnosis of non-metastatic cancer of any type (stage 0-3), including melanoma, colorectal, cervical, leukemia, lymphoma or breast cancer within the past 7 months
* Read and write English among their languages of choice
* Have ready access to a telephone
* Have a child 5-12 years old living at home who has been told their parent's cancer diagnosis
* The child is living at home and does not have learning challenges
* No prior malignancy is allowed except for adequately treated basal (or squamous cell) skin cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2014-04; Primary Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Recruitment and retention, monitored by tracking detailed recruitment spreadsheets | Up to 3 months
  Each referral source and method of referral will be monitored, including documenting reason for refusal. Four methods of recruitment will be monitored in order to know which method yields the highest enrollment: self-referral, provider referral, passive letter opt-in, and passive letter opt-out.
Dosage and fidelity, monitored for each intervention session using Performance Checklists | Up to 3 months
  Each audio-recorded intervention session will be reviewed against these checklists. Study participants' compliance with the in-session and at-home assignments will be monitored by the audio-recorded intervention sessions.
Acceptability of the program, assessed from interview data obtained from the Exit interview and the Swanson Caring Professional Scale | Up to 3 months
Rate of receipt of mailed materials both to participants and from participants | Up to 3 months
  Materials include signed consents, baseline data, and parent's educational materials.
Duration of phone intervention sessions | Up to 3 months
Rate of success in scheduling and completing intervention sessions by telephone | Up to 3 months
Quality of data on baseline and post-intervention measures | Up to 3 months
Short-term impact of the program, evaluated by comparing the change in pre- and post-test scores on the standardized questionnaires | Baseline up to 3 months
  Analysis of covariance (ANCOVA) will be used to test for significant differences between pre- and post-test scores, assuming the data meet the statistical assumptions. Baseline scores will serve as the covariate, along with empirical variables that are known to co-vary with parent and child functioning, e.g., length of time of diagnosis, type of medical treatment, adjuvant therapy, among others). Two-tailed tests of significance will be calculated, allowing us to evaluate any potential negative effects of the intervention.
Impact of the telephone-delivered compared to the in-person delivered program | Up to 3 months
  Linear mixed modeling will be used. Random effects models are based on Maximum Likelihood Estimation in which an iterative method estimates a trajectory for each study participant based on all available data for that participant supplemented by data obtained from the total sample.

CONTACTS AND LOCATIONS:
Overall Officials: Frances Lewis, Principal Investigator — Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium
Locations (11):
- United States (11):
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Tri-Cities Cancer Center, Kennewick, Washington
  - SCCA at EvergreenHealth, Kirkland, Washington
  - Skagit Valley Hospital, Mount Vernon, Washington
  - Olympic Medical Center, Port Angeles, Washington
  - Group Health Cooperative, Redmond, Washington
  - Fred Hutchinson Cancer Research Center/University of Washington Cancer Consortium, Seattle, Washington
  - Swedish Cancer Institute, Seattle, Washington
  - Multicare Health System, Tacoma, Washington
  - Wenatchee Valley Medical Center, Wenatchee, Washington